CLINICAL TRIAL: NCT05302466
Title: Additive Effects of Dental Bite Pads During Gymnastic Exercises for the Relief of Chronic Non-specific Neck Pain in Working Women and Men at a VDU Workplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ_2021
Record Dates: First submitted 2021-12-01; First posted 2022-03-31 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Chronic Neck Pain; TMD; Temporomandibular Dysfunction
Keywords: gymnastic; dental bite pad
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a monocentric, partially blinded, randomised clinical intervention study (RCT) in a parallel group design with participants from the Erlangen-Nuremberg area.
Who Masked: Outcomes Assessor
Masking Description: Computer-assisted block randomisation (stratification according to pain intensity) is carried out by an independent statistician. The blinding of the study refers to the measurement assistants who do not know/are not allowed to ask about the respective status of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gymnastic (control group) (Active Comparator): "usual care" home gymnastics programme for 12 weeks, which consists of three different 3-minute sequences to be performed daily.
  Interventions: Other: gymnastics only
- gymnastic plus dental bite pads (intervention group) (Experimental): Identical home gymnastics programme for 12 weeks, which consists of three different 3-minute sequences to be performed daily plus dental bite pads during exercise. The dental bite pads are placed on the back molars of the lower jaw and remain in this position in the mouth for 3 minutes during the exercise.
  Interventions: Device: gymnastics plus silicon dental bite pad

INTERVENTIONS:
Device: gymnastics plus silicon dental bite pad — Gymnastics (see below) plus dental bite pads. The dental bite pads TJ Motion (BELY Balance GmbH & Co. KG, Weisendorf, Germany) are made of medical silicone. Accordingly, they are BPA- and latex-free, odourless, tasteless and dimensionally stable. The splints are placed on the back molars of the lower jaw and remain in this position in the mouth for 3 minutes during the exercise. After use, the splints are rinsed with water and placed dry in the corresponding storage box.
  Other Names: TJ Motion
  Arms: gymnastic plus dental bite pads (intervention group)
Other: gymnastics only — Gymnastics, which are completed daily (7x/week), each consist of three to six exercises and have a total duration of three minutes. The gymnastic programme contain low-intensity exercises from functional gymnastic or physiotherapy.
  Other Names: exercise
  Arms: gymnastic (control group)

SUMMARY:
The study which includes 52 participants suffering from chronic neck pain, determines additional effects of dental bite pads on neck pain and function when performing a 3-month gymnastics programme.

DETAILED DESCRIPTION:
Chronic neck pain is a common health problem in our society. Targeted gymnastic exercises have a high priority in the context of therapy and have shown positive effects on the symptoms in studies. In the past, direct connections between the temporomandibular joint and complaints of the musculoskeletal system, especially of the shoulder-neck region, have been researched, which are based on neuroanatomical (nerves) and myofascial (muscle-fascia) connections. Against the background of current study results, consideration of these findings could be promising in the therapy of neck pain. A new approach tries to positively influence tension and discomfort in the neck area by changing the position of the temporomandibular joints using dental bite pads. In the planned study, the researchers are specifically investigating the question of the extent to which the placement of dental bite pads (made of silicone) in the molar region during the performance of gymnastic exercises can increase the effect of the exercises on neck pain and the associated restrictions on function and quality of life.

The aim of the present project is specifically to record the effect of a 3-month gymnastics programme and a possible additional effect of dental bite pads. In the study, 52 working women and men with a sedentary job at a computer workstation aged 30-65 years are included and randomly divided into two groups. Both groups will perform a specific video-animated exercise programme for 3 minutes 3 times a day over a period of 3 months with the main focus on the shoulder-neck region. One group positions a silicone dental bite pad (TJ Motion; BELY Balance GmbH & Co. KG, Weisendorf, Germany) on the right and left side of the molar region during the exercise.

Before the intervention, after 6 weeks and after a further 6 weeks of follow-up, pain and function in the neck area are assessed by questionnaire. At baseline and follow-up, functional tests of spinal and jaw mobility are also performed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 30-65 LJ
* Chronic non-specific neck pain [4] (at least for 3 months, pain intensity ≥2 (NRS) on at least 50% of days).
* Sedentary work, VDU work

Exclusion Criteria:

* Specific neck pain (e.g. herniated disc, spinal stenosis, etc.)
* Cervical spine-related neuronal symptoms (paresthesia, brachialgia, paresis)
* Continuous pain medication
* Concurrent other therapy to influence neck pain
* Absence ≥ 2 weeks during the intervention period
* Regular sports training (≥ 60min/week) in the last 6 months

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Neck pain (NRS) | Baseline, 6 Weeks, 12 Weeks
  Neck pain. The numerical rating scale (NRS) is a one-dimensional pain scale with which patients can quantify their subjectively felt pain. To do this, the patient is asked to assign their pain to a scale of 0-10. "10" stands for "strongest pain imaginable", "0" for "no pain". The recording is done every evening via a pain diary, in each case for one week, before the start of the intervention and in the 6th and 12th week of the intervention. The pain intensity as the primary endpoint is defined as the mean value over one week.

SECONDARY OUTCOMES:
Mobility of the cervical spine (range of motion (ROM)) | Baseline, 12 Weeks
  Sensor-based digital recording of flexion, extension, rotation, lateral flexion during active performance in a seated position (Mobeefit SportMed A.G. SA, Echternach, Luxembourg)
kyphosis angle | Baseline, 12 Weeks
  Posture (sagittal curvature / kyphosis angle (kyphometer n. Debrunner) in standing position
Shoulder mobility | Baseline, 12 Weeks
  End grade active flexion in sitting position (measurement bilaterally synchronous with goniometer))
TMD symptoms (questionnaires) | Baseline, 12 Weeks
  TMD Pain Screener, German version DC/TMD Symptom Questionnaire, German version Functional diagnostics of the temporomandibular joint

CONTACTS AND LOCATIONS:
Overall Officials: Simon von Stengel, Study Chair — University Erlangen-Nuremberg; Sebastian Willert, Principal Investigator — University Erlangen-Nuremberg; Wolfgang Kemmler, PhD, Study Director — University Erlangen-Nuremberg
Locations (1):
- Institute of medical physics, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No